CLINICAL TRIAL: NCT03633591
Title: A Phase 1, Single-Part, 6-Period, Sequential, Non-Randomized, Open-Label Study Designed to Evaluate the Pharmacokinetic Profile of Tolcapone Following Administration of Modified Release Prototype Formulations and an Experimental Divided Dose Regimen in Healthy Subjects
Brief Title: A Study Assessing the Safety and Pharmacokinetic Profile of Modified Release Formulations of Tolcapone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corino Therapeutics, Inc. (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TOLC101MR; 2017-003070-13 (EudraCT Number)
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tolcapone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified Release Prototypes of Tolcapone (Experimental)
  Interventions: Drug: Tolcapone; Drug: Tolcapone Modified Release Prototype; Drug: Tolcapone Divided Dose

INTERVENTIONS:
Drug: Tolcapone — Multiple doses of tolcapone tablets in the fasted state
  Other Names: Tasmar
Drug: Tolcapone Modified Release Prototype — A single dose of tolcapone modified release prototype in the fasted state
Drug: Tolcapone Divided Dose — Tolcapone (suspension) in equal divided doses in the fasted state
Drug: Tolcapone Modified Release Prototype — A single dose of tolcapone modified release prototype (optionally two doses or fed state of prior MR prototype)

SUMMARY:
The purpose of this study is to assess the pharmacokinetic profiles of tolcapone in healthy subjects after administration of one or two oral doses of multiple modified release prototype formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Age 18 to 65 years of age at the time of signing informed consent
* Body mass index (BMI) of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months prior to first dose.
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
* Subjects who have previously been enrolled in this study.
* History of any drug or alcohol abuse in the past 2 years.
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Females of childbearing potential who are pregnant or lactating
* Subjects who do not have suitable veins for multiple venepunctures / cannulation as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the investigator
* Hemoglobin below the lower limit of normal
* ALT or AST outside the normal reference range at screening or admission.
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of clinically significant cardiovascular, neurological, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder, as judged by the investigator
* Subjects with a history of cholecystectomy or gall stones
* Serious adverse reaction or serious hypersensitivity to any drug, the formulation excipients, or lactose intolerance
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator.
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before IMP administration.
* Contraindication for Tasmar®
* Failure to satisfy the investigator of fitness to participate for any other reason

NOTE: Other inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment: Time to maximum concentration (Tmax) | Pre-dose to 24 hours post-dose
  Time to maximum concentration (Tmax)
Pharmacokinetic Assessment: Maximum observed concentration (Cmax) | Pre-dose to 24 hours post-dose
  Maximum observed concentration (Cmax)
Pharmacokinetic Assessment: Area under the curve (AUC) | Pre-dose to 24 hours post-dose
  Area under the curve (AUC)
Pharmacokinetic Assessment: Plasma half-life (t1/2) | Pre-dose to 24 hours post-dose
  Plasma half-life (t1/2)
Pharmacokinetic Assessment: Relative bioavailability (Frel) | Pre-dose to 24 hours post-dose
  Relative bioavailability (Frel)

SECONDARY OUTCOMES:
Pharmacokinetic Assessment of 3-O-Methyltolcapone: Time to maximum concentration (Tmax) | Pre-dose to 24 hours post-dose
  Time to maximum concentration (Tmax)
Pharmacokinetic Assessment of 3-O-Methyltolcapone: Maximum observed concentration (Cmax) | Pre-dose to 24 hours post-dose
  Maximum observed concentration (Cmax)
Pharmacokinetic Assessment of 3-O-Methyltolcapone: Area under the curve (AUC) | Pre-dose to 24 hours post-dose
  Area under the curve (AUC)
Pharmacokinetic Assessment of 3-O-Methyltolcapone: Plasma half-life (t1/2) | Pre-dose to 24 hours post-dose
  Plasma half-life (t1/2)
Pharmacokinetic Assessment of 3-O-Methyltolcapone: Relative Bioavailability (Frel) | Pre-dose to 24 hours post-dose
  Relative Bioavailability (Frel)
Number of subjects reporting treatment-related Adverse Events (AEs) | Screening to 10 days following last dose
  Abnormalities in safety laboratory tests, vital signs, electrocardiogram, physical examination that meet the protocol definition will be captured as AEs

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No